CLINICAL TRIAL: NCT06815120
Title: Two Single Arm, Multicentre Unblinded First-in-human Trials Investigating a Novel Ureteric Stent to Determine the Reduction of Encrustation, Biofilm Deposition and Complications Compared to a Conventional JJ Stent
Brief Title: A Novel Ureteric Stent in Kidney Stone Patients and Oncology Patients Compared to a Conventional JJ Stent
Acronym: CASSETTE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: University Hospital Southampton NHS Foundation Trust (Other); National Institute for Health Research, United Kingdom (Other Government); University College London Hospitals (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 63246
Record Dates: First submitted 2024-12-04; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Catheter Blockage; Oncology; Kidney Stone
MeSH Terms: conditions — Neoplasms; Kidney Calculi

STUDY DESIGN:
Intervention Model Description: Two single arm, multicentre unblinded first-in-human trials, including 2 phases and a qualitative substudy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Kidney Stone cohort (Experimental): Experimental ureteric stent with specially shaped side-holes that prevent stagnation points (i.e., areas of low flow that cause particles to settle and E&B)
  Interventions: Device: Experimental ureteric stent with specially shaped side-holes that prevent stagnation points (i.e., areas of low flow that cause particles to settle and E&B); Other: Qualitative interview
- Oncology cohort (Experimental): Experimental ureteric stent with specially shaped side-holes that prevent stagnation points (i.e., areas of low flow that cause particles to settle and E&B)
  Interventions: Device: Experimental ureteric stent with specially shaped side-holes that prevent stagnation points (i.e., areas of low flow that cause particles to settle and E&B); Other: Qualitative interview

INTERVENTIONS:
Device: Experimental ureteric stent with specially shaped side-holes that prevent stagnation points (i.e., areas of low flow that cause particles to settle and E&B) — Kidney stone patients and Oncology patients admitted to either the University Hospital Southampton (UHS) or University College London Hospital (UCLH) for management of kidney stones or for the management of urine drainage in ureter will have a novel ureteric stent instead of their planned conventional stent. The novel stent will be removed after 4 weeks (kidney stone patients) or 25 weeks (oncology patients). Recruitment to the cohort of oncology patients will only commence once the results for kidney stones patients have been reviewed.
Other: Qualitative interview — Kidney stone patients, Oncology patients and doctors will be interviewed about their experience of having a stent, or their experience in managing patients with a stent.

SUMMARY:
Urological stents and catheters often lead to inflammation, causing pain and infection in the urinary tract. Moreover, 80% of stents are associated with pain, negatively impacting on QoL and mental health. Offering novel designs with significantly lower E&B leads to a reduction in UTIs and improves QoL. Reducing hospital admissions (from 3 to 1 per patient, annually) would free >100,000 bed-nights, allowing the elderly to regain independence. Our proposed research could have a significant impact towards fulfilling the 'healthy-ageing' Grand Challenge. Additionally, the novel stent reduces prevalence of infections and therefore, of antibiotic prescriptions contributing to the Global AMR challenge.

DETAILED DESCRIPTION:
Ureteric stents and catheters are deployed clinically as temporary measures to restore urinary drainage, in patients with kidney stones, tumours and strictures. Prevalence of these increases with age. Device-associated encrustation-and-biofilm-formation (E&B) are key complications, leading to urinary-tract-infections (UTIs) in >90% of stents, causing stent blockage and favouring development of antibiotic resistance.

UTIs are a significant cause of morbidity, especially among the elderly population, with 4,835 deaths in England and Wales reported in 2012. The National Institute for Health Research reported that 1-3% of all primary care consultations concern UTI-related symptoms, leading to 13.7% of antibiotic prescriptions globally. The report also revealed that >92m people globally are diagnosed with UTIs annually.

Urological-device-associated infections significantly compromise patient' quality of life and the effectiveness of services, imposing a £2.5b annual burden on the NHS. Patients' exposure to hospital environment and general anaesthetic use impact on Quality-of-Life (QoL), resulting in unnecessary hospital bed-nights. We have developed a novel urological stent associated with significantly reduced particle deposition , potentially extending the stent's lifetime, resulting in reduced hospitalisation and improved QoL.

Urological stents and catheters often lead to inflammation, causing pain and infection in the urinary tract. Moreover, 80% of stents are associated with pain, negatively impacting on QoL and mental health. Offering novel designs with significantly lower E&B leads to a reduction in UTIs and improves QoL. Reducing hospital admissions (from 3 to 1 per patient, annually) would free >100,000 bed-nights, allowing the elderly to regain independence. Our proposed research could have a significant impact towards fulfilling the 'healthy-ageing' Grand Challenge. Additionally, the novel stent reduces prevalence of infections and therefore, of antibiotic prescriptions contributing to the Global AMR challenge.

Considering only onco-urological patients, >30,000 stents are inserted every year across 200 NHS units. Due to stent failures, each patient undergoes 3 to 6 replacements, resulting in >90,000 stent replacements. Under the current tariff-based system, hospitals are paid for each intervention, costing the NHS >£3,500, bringing the total cost of replacements to ~£315m annually. Unnecessary replacements increase the number of bed-nights and use of anaesthetics. A longer-lasting stent means that each patient comes to the hospital ideally only once, reducing their exposure to the hospital environment and anaesthetic-associated risks. Additionally, under the current model hospitals would improve their quality of service and save at least 2 bed-nights per patient. The NHS is moving towards a "block contract" model, meaning that hospitals will receive a lump sum for the year and they'll regularly monitor budgets and improve cost efficiency where possible. Improved stents will allow the same urology budget to deliver more healthcare, reducing theatre time for stent insertion-and-replacement. Our innovative stent design offers a potential annual saving of >£210m for the NHS, allowing hospitals to reallocate their resources. Today E&B is still a major determinant of stent failure and associated side effects. We aim to address this challenge through our novel stent, and if equivalent safety and improved efficacy are demonstrated, anticipate market launch via third-party suppliers 2-3 years post project.

Solutions to break this pathway (stent presence >> inflammation, pain and infection) have been developed, including materials (e.g. metallic alloys, polymers, biodegradable and drug-eluting materials), coatings (e.g. heparin, chitosan, hydrogel, carbon) and shapes (e.g. double-J, loop, mesh, string, expandable) to improve the efficacy and safety of stents. Despite all these advances, there is still a significant prevalence of E&B. This is also due to the lack of studies correlating fluid dynamic metrics with deposition of particles causing E&B. The lead applicant's PhD investigated the mechanisms of particle deposition in urological stents, and successfully determined fluid dynamic parameters governing particle deposition on ureteric stents and catheters. His research led to developing a stent with specially shaped side-holes that prevent stagnation points (i.e., areas of low flow that cause particles to settle and E&B). These developments demonstrated >80% reduction in particle deposition at side-holes, in-vitro. Their innovative architecture can be implemented on stents and catheters. The technology, including the stent design and manufacturing process, is protectable - Patent# WO2019048860A1, WIPO(PCT). These results were further validated in an animal study (6 pigs: 3 novel-design-stent vs 3 conventional-design-stent for a 4-weeks period) at Stone-Centre at Vancouver-General-Hospital (VGH), a centre of excellence in animal studies on urological products. The study (available upon request) concluded that the functionality of stents with novel side-holes is the same as that of standard stents in terms of safety. Specifically, the novel stent does not result in increased risk of irritation, inflammation and hydronephrosis. Furthermore, SEM/EDX imaging showed that the novel design decreased the build-up of particles on the stent surface. Thus, it demonstrated significant potential for the new side-hole configuration to change patterns of particle deposition on the stent's surface, decreasing encrustation

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or over
2. Ureteric stents clinically indicated either due to kidney stones or abdominal/pelvic cancers compressing ureters
3. Previous experience with ureteric stents
4. Awaiting insersion/replacement of stents
5. Ability to give consent
6. Ability to interact with study documentation
7. Sufficient English to complete study documentations and questionnaires

Exclusion Criteria:

1. Expected survival <4months
2. Unfit for stent insertion
3. Unable to comply with study processes Pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
To determine rates of stent failure | From enrolment to stent removal (4 weeks for Kidney cohort), (25 weeks for Oncology cohort)
  Outcome measure: Stent failure, defined as any of: a): a stent change earlier than planned (oncology only); b) need for additional surgical or radiological intervention; c): kidney failure (evidenced by acute kidney injury (AKI) on blood tests (eGFR or creatinine kidney function tests) and/or worsening hydronephrosis on imaging
  Summary method: Frequency and percentage of people experiencing any stent failure

SECONDARY OUTCOMES:
To assess extent of encrustation and biofilm (E&B) | From enrolment to stent removal (4 weeks for Kidney cohort), (25 weeks for Oncology cohort)
  Outcome measure:
  * Cell culturing (CFU counts per ml per bacterial microorganism)
  * Flow study (pressure value): A section of the retrieved stent will be used for flow study. The part will be placed into a larger diameter tube. DI water/Saline is injected using a pump into the inlet of the external tube and pressure sensor is connected to the inlet tube. Pressure readings will be captured per stent.
  * Dwell time
  Summary method:
  * Imaging (selected samples of stents will be examined using non-contact, non-destructive SEM (scanning-electron-microscopy) and/or episcopic-differential-interference-contrast (EDIC) microscopy allowing imaging of the surface with the biofilm in-situ and colonisation by bacteria - when needed)
  * Mean and standard deviation or median and quartiles of pressure readings
To determine whether the novel stent leads to better clinical outcomes | From enrolment to completion of patient questionnaires 2-3 weeks post surgery 2 (4 weeks for Kidney cohort), 2-3 weeks post surgery 2 (~25 weeks for Oncology cohort)
  Outcome measure:
  * Individual component of the primary outcome
  * Urinary symptoms
  * Infections
  Summary method:
  * As per primary outcome
  * Frequency and percentage of participants experiencing each symptom
  * Frequency and percentage of people with antibiotic
  * use, readmission, urosepsis, ITU, death; number of infections per unit of time stent is in use
To assess impact of the novel stent on quality of life | Within first month of stent removal for participants (4 weeks for Kidney cohort), (25 weeks for Oncology cohort)
  Outcome measure:
  Questionnaires at:
  * Baseline
  * While stent is in situ
  * Post-surgery
  Summary method:
  Appropriate descriptive summaries (e.g., median and quartiles) per timepoint
To understand patient experience in having the novel ureteric stent inserted and reason for participation in the trial | From enrolment to stent removal (4 weeks for Kidney cohort), (25 weeks for Oncology cohort)
  Outcome measure:
  30-45-minute Qualitative interviews with Oncology and Kidney stone cohorts
  Summary method:
  An inductive thematic analysis of interview transcripts

OTHER OUTCOMES:
To assess extent of encrustation and biofilm (E&B) | After surgery 2 for Kidney Stone cohort (4 weeks) and surgery 2 for Oncology patients (25 weeks)
  Outcome measure:
  Weight: Weighing stents after being removed from body, at the site (theatre room) and prior to packaging for delivery to the University laboratory
  Summary method:
  Mean and standard deviation or median and quartiles of weights pre- and post-insertion

CONTACTS AND LOCATIONS:
Overall Officials: Ali Mosayyebi, Principal Investigator — University of Southampton

IPD SHARING:
Plan to Share IPD: Undecided
To be decided

REFERENCES:
- [Background] Prattley S, Voss J, Cheung S, Geraghty R, Jones P, Somani BK. Ureteroscopy and stone treatment in the elderly (>/=70 years): prospective outcomes over 5- years with a review of literature. Int Braz J Urol. 2018 Jul-Aug;44(4):750-757. doi: 10.1590/S1677-5538.IBJU.2017.0516. PMID 29522293
- [Background] Heers H, Turney BW. Trends in urological stone disease: a 5-year update of hospital episode statistics. BJU Int. 2016 Nov;118(5):785-789. doi: 10.1111/bju.13520. Epub 2016 May 26. PMID 27128735
- [Background] Z. Chen, M. Prosperi, and V. Y. Bird, "Prevalence of kidney stones in the USA: The National Health and Nutrition Evaluation Survey," J Clin Urol, vol. 12, no. 4, pp. 296-302, Jul. 2019, doi: 10.1177/2051415818813820
- [Background] C. R. UK, "Cancer incidence by age," 2020. https://www.cancerresearchuk.org/health-professional/cancer-statistics/incidence/age#heading-Zero (accessed Apr. 11, 2021)
- [Background] Kehinde EO, Rotimi VO, Al-Hunayan A, Abdul-Halim H, Boland F, Al-Awadi KA. Bacteriology of urinary tract infection associated with indwelling J ureteral stents. J Endourol. 2004 Nov;18(9):891-6. doi: 10.1089/end.2004.18.891. PMID 15659928
- [Background] S. T. Thomas, C. Heneghan, C. P. Price, A. van den Bruel, and A. Plüddemann, "Point-of-care testing for urinary tract infections - NIHR Community Healthcare MIC," NIHR, Jun. 2016. https://www.community.healthcare.mic.nihr.ac.uk/reports-and-resources/horizon-scanning-reports/point-of-care-testing-for-urinary-tract-infections (accessed Feb. 01, 2023)
- [Background] Zumstein V, Betschart P, Albrich WC, Buhmann MT, Ren Q, Schmid HP, Abt D. Biofilm formation on ureteral stents - Incidence, clinical impact, and prevention. Swiss Med Wkly. 2017 Feb 3;147:w14408. doi: 10.4414/smw.2017.14408. eCollection 2017. PMID 28165539
- [Background] Feneley RC, Hopley IB, Wells PN. Urinary catheters: history, current status, adverse events and research agenda. J Med Eng Technol. 2015;39(8):459-70. doi: 10.3109/03091902.2015.1085600. Epub 2015 Sep 18. PMID 26383168
- [Background] Joshi HB, Stainthorpe A, MacDonagh RP, Keeley FX Jr, Timoney AG, Barry MJ. Indwelling ureteral stents: evaluation of symptoms, quality of life and utility. J Urol. 2003 Mar;169(3):1065-9; discussion 1069. doi: 10.1097/01.ju.0000048980.33855.90. PMID 12576847
- [Background] Ramachandra M, Mosayyebi A, Carugo D, Somani BK. Strategies to Improve Patient Outcomes and QOL: Current Complications of the Design and Placements of Ureteric Stents. Res Rep Urol. 2020 Jul 31;12:303-314. doi: 10.2147/RRU.S233981. eCollection 2020. PMID 32802807
- [Background] Mosayyebi A, Manes C, Carugo D, Somani BK. Advances in Ureteral Stent Design and Materials. Curr Urol Rep. 2018 Apr 10;19(5):35. doi: 10.1007/s11934-018-0779-y. PMID 29637309
- [Background] Mosayyebi A, Vijayakumar A, Yue QY, Bres-Niewada E, Manes C, Carugo D, Somani BK. Engineering solutions to ureteral stents: material, coating and design. Cent European J Urol. 2017;70(3):270-274. doi: 10.5173/ceju.2017.1520. Epub 2017 Aug 28. PMID 29104790
- [Background] Liatsikos EN, Kallidonis P, Kyriazis I, Karnabatidis D, Tsamandas A, Sakellaropoulos G, Flaris N, Rigopoulos C, Toronidis C, Efthimiou I, Filos K, Siablis D, Perimenis P. Metallic double pigtail ureteral stent usage during extracorporeal shock wave lithotripsy in the swine model: is there any effect on the ureter? J Endourol. 2009 Apr;23(4):685-91. doi: 10.1089/end.2008.0569. PMID 19335328
- [Background] S. Zheng et al., "Quantitative Evaluation of Encrustations in Double-J Ureteral Stents With Micro-Computed Tomography and Semantic Segmentation," Frontiers in Urology, vol. 2, 2022, [Online]. Available: https://www.frontiersin.org/articles/10.3389/fruro.2022.836563
- [Background] Tomer N, Garden E, Small A, Palese M. Ureteral Stent Encrustation: Epidemiology, Pathophysiology, Management and Current Technology. J Urol. 2021 Jan;205(1):68-77. doi: 10.1097/JU.0000000000001343. Epub 2020 Aug 28. PMID 32856981
- [Background] Mosayyebi A, Lange D, Yann Yue Q, Somani BK, Zhang X, Manes C, Carugo D. Reducing deposition of encrustation in ureteric stents by changing the stent architecture: A microfluidic-based investigation. Biomicrofluidics. 2019 Jan 4;13(1):014101. doi: 10.1063/1.5059370. eCollection 2019 Jan. PMID 30867872
- [Background] Mosayyebi A, Yue QY, Somani BK, Zhang X, Manes C, Carugo D. Particle Accumulation in Ureteral Stents Is Governed by Fluid Dynamics: In Vitro Study Using a "Stent-on-Chip" Model. J Endourol. 2018 Jul;32(7):639-646. doi: 10.1089/end.2017.0946. Epub 2018 Jun 12. PMID 29699424
- [Background] Rosenthal R, Schafer J, Briel M, Bucher HC, Oertli D, Dell-Kuster S. How to write a surgical clinical research protocol: literature review and practical guide. Am J Surg. 2014 Feb;207(2):299-312. doi: 10.1016/j.amjsurg.2013.07.039. Epub 2013 Oct 26. PMID 24262932
- [Background] Newcombe RG. Two-sided confidence intervals for the single proportion: comparison of seven methods. Stat Med. 1998 Apr 30;17(8):857-72. doi: 10.1002/(sici)1097-0258(19980430)17:83.0.co;2-e. PMID 9595616
- See also: NHS, "Overview - Hydronephrosis," NHS website, 2018 — http://www.nhs.uk/conditions/hydronephrosis/